CLINICAL TRIAL: NCT01029262
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study To Compare The Efficacy And Safety of Lenalidomide (Revlimid®) Versus Placebo In Subjects With Transufsion-Dependent Anemia Due to IPSS Low Or Imtermidate-1 Risk Myelodysplastic Syndromes Without Deletion 5Q(31) And Unresponsive Or Refractory To Erthropoiesis-Stimulating Agents
Brief Title: A Study of Lenalidomide Versus Placebo in Subjects With Transfusion Dependent Anemia in Lower Risk Myelodysplastic Syndrome (MDS) Without Del 5q
Acronym: MDS-005
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-MDS-005
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Anemia
Keywords: Myelodysplastic Syndromes; MDS; transfusion dependent anemia; Erythropoiesis stimulating agents; non-del 5q
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm #1 - Lenalidomide plus placebo (Experimental): Lenalidomide 10 mg by mouth (PO) daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 60 mL/min for at least 168 days until disease progression, intolerable side effects or withdrawal of consent. Lenalidomide 5 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 40 and < 60 mL/min.
  Interventions: Drug: Lenalidomide
- Arm #2 - placebo (Placebo Comparator): Three placebo capsules once daily for at least 168 days until disease progression occurred, intolerable side effects or withdrawal of consent.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lenalidomide — One 10 mg Lenalidomide capsule + 2 placebo capsules or (3 placebo capsules) once daily for subjects with a creatinine clearance ≥ 60 mL/min. Alternatively-one 5 mg Lenalidomide capsule + 2 placebo capsules (or 3 placebo capsules) once daily for subjects with a creatinine clearance between 40 and 60 mL/min. Subjects may take study drug for at least 168 days unless there are intolerable side effects or disease progresses. Subjects may continue study drug beyond 168 days if they have an erythroid response (increase in their hemoglobin levels and fewer transfusions administered than before starting study drug)
  Other Names: Revlimid; CC-5013
  Arms: Arm #1 - Lenalidomide plus placebo
Other: Placebo — 3 placebo capsules once daily. Subjects may take study drug for at least 168 days unless there are intolerable side effects or disease progresses. Subjects may continue study drug beyond 168 days if they have an erythroid response (increase in their hemoglobin levels and fewer transfusions administered than before starting study drug)
  Arms: Arm #2 - placebo

SUMMARY:
The purpose of this study is to investigate whether lenalidomide would reduce the number of red blood cell transfusions (RBC) needed in anemic (RBC transfusion-dependent) participants with low or intermediate-1 risk MDS without a deletion 5q chromosome abnormality. The study also investigated the safety of lenalidomide use in these participants. Two-thirds of the participants received oral lenalidomide and one-third of the participants received oral placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of low or intermediate-1 risk Myelodysplastic (MDS) with any chromosome karyotype except del 5q[31]
* Anemia that requires red blood cell transfusions
* Resistant to erythropoiesis stimulating agents (ESAs) or blood erythropoietin level > 500 mU/mL
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2
* Must agree to follow pregnancy precautions as required by the protocol.
* Must agree to receive counseling related to teratogenic and other risks of lenalidomide
* Must agree not to donate blood or semen
* Must be willing to consent to two or more bone marrow aspirate procedures to be completed during study

Exclusion Criteria:

* Subjects previously receiving immunomodulating or immunosuppressive agents, or epigenetic or deoxyribonucleic acid (DNA) modulation agents
* Allergic reaction to thalidomide
* Renal insufficiency creatinine clearance (CrC1)<40 mL/min by Cockcroft-Gault method)
* Prior history of cancer, other than MDS, unless the subject has been free of the disease for ≥ 5 years. (Basal cell carcinoma of the skin, carcinoma in situ of the cervix, or stage Tumor (T) 1a or T1b prostate cancer is allowed)
* Absolute neutrophil count (ANC) < 500/uL
* Platelets < 50,000/uL
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3X upper limit of normal
* Uncontrolled hyperthyroidism or hypothyroidism
* Significant neuropathy
* Prior stem cell transplantation
* Anemia due to reasons other than MDS
* History of deep venous thrombosis (DVT) or pulmonary embolus (PE) within past 3 years
* Significant active cardiac disease within the past 6 months
* Known Human Immunodeficiency Virus (HIV) infection; known Hepatitis C infection or active Hepatitis B infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2010-01-26 (Actual); Primary Completion 2013-03-17 (Actual); Study Completion 2018-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Hoenekopp, MD, Study Director — Celgene Corporation
Locations (99):
- United States (7):
  - University of California at Los Angeles, Los Angeles, California
  - Southern Illinois Hematology Oncology, Centralia, Illinois
  - Dartmouth Hitchcock Medical Center Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Adelaide Hospital Institute of Medical and Veterinary Science, Adelaide, South Australia
  - Princess Alexandra Hospital, Woolloongabba
- Austria (5):
  - Medizinische Universitat Innsbruck, Innsbruck
  - Krankenhaus der Elisabethinen Linz, I Interne Abteilung, Linz
  - Universitatsklinik fur Innere Medizin Salzburg, Salzburg
  - Wiener Gebietskrankenkasse-Hanusch-Krankenhaus, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Weis
- Belgium (7):
  - AZ St-Jan Brugge Oostende AV, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Centre Hospitalier Universitaire de Liege, Liège
  - Center Hospitalier Universitaire Ambroise Pare, Mons
  - Cliniques Universitaires UCL de Mont-Godine, Namur
- Canada (8):
  - Tom Baker Cancer Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Cancer Care Manitoba, Winnepeg, Manitoba
  - Sunnybrook Regional Cancer Center, Toronto, Ontario
  - Princess Margaret Hospital and University of Toronto, Toronto, Ontario
  - Maisonneuve Rosemont, Montreal, Quebec
  - McGill University, Dept. Oncology Clinical Research Program, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Ustav hematologie a krevni transfuze, Prague
  - Vseobecna Fakultni Nemocnice v Praze, Prague
- France (6):
  - CHU d'Angers, Angers
  - Hopital Avicenne, Bobigny
  - Hopital A. Michallon, La Tronche
  - CHRU de Lille-Hopital Claude Huriez Service des Maladies du Sang, Lille
  - Institut Paoli-Calmettes, Marseille
  - Groupe hospitalier Cochin Saint-Vincent de Paul, Paris
- Germany (9):
  - Universitat zu Koln, Cologne
  - BAG Freiberg-Richter, Jacobash, Illmer, Wolf, Dresden
  - Sankt Johannes Hospital Duisburg, Duisberg
  - Universitätsklinikum Düsseldorf, Düesseldorf
  - Marien Hospital, Düsseldorf
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Mannheim der Universitat Heidelberg, Heidelberg
  - Universitatsklinikum Mannheim, Mannheim
  - TU München - Klinikum rechts der Isar, München
- Israel (3):
  - Rabin Medical Center, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (12):
  - Az. Osp. SS.Antonio e Biagio - SC Ematologia, Alessandria
  - A.O.U. di Bologna Policlinico S.Orsola-Malpighi, Bologna
  - P.O. Ospedale Roberto Binaghi (UNI CA/ASL 8), Cagliari
  - Azienda Ospedaliero-Universitaria di Cagliari, Cagliari
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Azienda Ospedaliera Cardarelli, Naples
  - AOU San Luigi Gonzaga, Orbassano
  - IRCCS Centro di Riferimento Oncologico di Basilicata di Rionero in Vulture, Rionero in Vulture
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
  - Azienda Policlinico Umberto I, Universita La Sapienzadi Roma, Roma
  - Policlinico Agostino Gemelli - Istituto di Ematologia, Roma
  - Policlinico Univeristario di Udine, Udine
- Japan (11):
  - Hiroshima University Hospital, Hiroshima
  - Tokai University School of Medicine, Isehara City, Kanagawa
  - Kameda General Hospital, Kamogawa
  - Kanazawa University Hospital, Kanazawa
  - Nagasaki Unversity Hospital, Nagasaki
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Osaka Red Cross Hospital, Osaka
  - Tohoku University Hospital, Sendai
  - Japanese Red Cross Medical Center, Shibuya City
  - Jichi Medical University Hospital, Shimotsuke
  - Kanto Medical Center NTT EC, Shinagawa City
- Poland (3):
  - Katedra i Klinika Hematologii i Transplantacji Szpiku - SLASKIEGO UNIWERSYTETU MEDYCZNEGO, Gdansk
  - Uniwersytet Medyczny w Lodzi, Lodz
  - Instytut Hematologii i Transfuzjologii, Klinika Hematologii, Warsaw
- Portugal (3):
  - Hospitais da Universidade de Coimbra, Coimbra
  - Instituto Portugues de Oncologia de Lisboa, Lisbon
  - Hospital Geral de Santo Antonio, Porto
- Spain (7):
  - Hospital Clinic Provincial de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario La Fe, Valencia
- Turkey (Türkiye) (4):
  - Gazi Universitesi Tip Fakltesi, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Istanbul Universitesi Istanbul, Istanbul
  - Dokuz Eylul Universitesi Tip Faiultesi, Izimir
- United Kingdom (7):
  - Royal Bournemouth Hospital, Bournemouth
  - University Hospital of Wales, Cardiff
  - Saint James University Hospital, Leeds
  - Barts Cancer Institute, Queen Mary University of London, Charterhouse Square, London
  - King's College Hospital, London
  - Christie Hospital, Manchester
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Result] Santini V, Almeida A, Giagounidis A, Gropper S, Jonasova A, Vey N, Mufti GJ, Buckstein R, Mittelman M, Platzbecker U, Shpilberg O, Ram R, Del Canizo C, Gattermann N, Ozawa K, Risueno A, MacBeth KJ, Zhong J, Seguy F, Hoenekopp A, Beach CL, Fenaux P. Randomized Phase III Study of Lenalidomide Versus Placebo in RBC Transfusion-Dependent Patients With Lower-Risk Non-del(5q) Myelodysplastic Syndromes and Ineligible for or Refractory to Erythropoiesis-Stimulating Agents. J Clin Oncol. 2016 Sep 1;34(25):2988-96. doi: 10.1200/JCO.2015.66.0118. Epub 2016 Jun 27. PMID 27354480
- [Derived] Santini V, Almeida A, Giagounidis A, Skikne B, Beach CL, Weaver J, Tu N, Fenaux P. Achievement of red blood cell transfusion independence in red blood cell transfusion-dependent patients with lower-risk non-del(5q) myelodysplastic syndromes correlates with serum erythropoietin levels. Leuk Lymphoma. 2020 Jun;61(6):1475-1483. doi: 10.1080/10428194.2020.1719088. Epub 2020 Feb 17. PMID 32064987
- [Derived] Almeida A, Fenaux P, Garcia-Manero G, Goldberg SL, Gropper S, Jonasova A, Vey N, Castaneda C, Zhong J, Beach CL, Santini V. Safety profile of lenalidomide in patients with lower-risk myelodysplastic syndromes without del(5q): results of a phase 3 trial. Leuk Lymphoma. 2018 Sep;59(9):2135-2143. doi: 10.1080/10428194.2017.1421758. Epub 2018 Jan 11. PMID 29322849

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 239 participants were randomized at sites located in Europe (185), North America (24), Asia/Pacific (13) and the Middle East (17).
Pre-assignment Details: Participants must have had transfusion-dependent anemia defined as having an average transfusion need of at least 2 units of packed red blood cells (pRBCs) per 28 days during the 112 days preceding randomization; No consecutive 56-day period that was RBC-transfusion-free during the 112 days preceding randomization; hemoglobin levels ≤ 9.5 g/dL.
Groups:
- Placebo: Participants received 3 placebo capsules by mouth (PO) daily (QD) for at least 168 days until disease progression occurred, intolerable side effects or withdrawal of consent.
- Lenalidomide: Participants received lenalidomide 10 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 60 mL/min for at least 168 days until disease progression, intolerable side effects or withdrawal of consent.
  Participants received lenalidomide 5 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 40 and < 60 mL/min.
Period: Overall Study
Arm/Group | Placebo | Lenalidomide
Started | 79 | 160
Completed | 0 | 0
Not Completed | 79 | 160
Not completed — Adverse Event | 9 | 52
Not completed — Lack of therapeutic effect | 57 | 76
Not completed — Withdrawal by Subject | 10 | 17
Not completed — Protocol Violation | 2 | 3
Not completed — Miscellaneous | 1 | 9
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population includes all participants who were randomized.
Groups:
- Placebo: Participants received 3 placebo capsules by mouth daily for at least 168 days until disease progression occurred, intolerable side effects or withdrawal of consent.
- Lenalidomide: Participants receieved lenalidomide 10 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 60 mL/min for at least 168 days until disease progression, intolerable side effects or withdrawal of consent.
  Lenalidomide 5 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 40 and < 60 mL/min.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lenalidomide | Total
Number analyzed (Participants) | 79 | 160 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (8.26) | 70.0 (8.19) | 69.6 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 52 | 77
  Male | 54 | 108 | 162
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 0 | 2 | 2
  White | 69 | 133 | 202
  Japanese | 4 | 8 | 12
  Race Not Disclosed | 4 | 15 | 19
  Other | 1 | 1 | 2
Packed RBC (pRBC) Transfusion Burden [Mean (Standard Deviation); unit: pRBC units/28 days] — The baseline transfusion burden is the average number of RBC units/28 days during the 112 days prior to randomization.
  pRBC units/28 days | 3.4 (1.37) | 3.4 (1.23) | 3.4 (1.28)
International Prognostic Scoring System (IPSS) Investigator Determined [Count of Participants; unit: Participants] — The Myelodysplastic Syndrome (MDS) IPSS score assesses the severity of MDS based on 3 prognostic factors each assigned a score: the percentage of bone marrow blasts, chromosome changes in the marrow cells (karyotype) and the presence of one or more low blood cell counts (cytopenias). The IPSS score is the sum of the bone marrow blast + karyotype + cytopenia score and ranges from 0 (low risk) to 3.5 (high risk). Prognosis is categorized as Low risk (score = 0), Intermediate-1 (score 0.5 to 1.0), Intermediate-2 (score 1.5 to 2.0) or High risk (score ≥ 2.5).
  Participants
    Low | 30 | 85 | 115
    Intermediate 1 | 49 | 75 | 124
World Health Organization Classification 2008 of MDS by Central Review [Count of Participants; unit: Participants] — The World Health Organization (WHO) 2008 classification recognizes eight subtypes of MDS that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts (i.e., erythroid precursors with iron deposits surrounding the nucleus), presence of a monocytosis or a deletion 5q.
  Participants
    Refractory anemia (RA) | 1 | 1 | 2
    Refractory cytopenia unilineage dysplasia (RCUD) | 0 | 5 | 5
    RA with ringed sideroblasts (RARS) | 7 | 12 | 19
    Refractory cytopenia multilineage dysplasia (RCMD) | 59 | 115 | 174
    Refractory anemia with excess blasts-1 (RAEB-1) | 12 | 27 | 39
Prior Erythropoiesis-stimulating Agent (ESA) Treatment [Count of Participants; unit: Participants] — Erythropoiesis-stimulating agents (ESA) are similar to the cytokine (erythropoietin) that stimulates red blood cell production (erythropoieisis). ESAs, structurally and biologically, are similar to naturally occurring protein erythropoietin. ESAs are used to maintain hemoglobin at the lowest level that both minimizes transfusions and best meets a person's needs
  Participants
    Yes | 63 | 125 | 188
    No | 16 | 35 | 51
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 8.7 (1.37) | 8.7 (1.23) | 8.7 (1.28)
Gene Expression Signature [Count of Participants; unit: Participants] — A prespecified subgroup of participants with an erythroid differentiation gene expression signature predictive of lenalidomide response
  Participants | 3 | 14 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Red Blood Cell (RBC) Transfusion Independence for ≥ 56 Days as Determined by an Independent Review Committee (IRC)
Description: The percentage of participants who achieved the 56-day RBC transfusion independent (TI) response was defined as the absence of any RBC transfusions during any consecutive "rolling" 56-day interval within the double-blind treatment phase (ie, Days 2 (Day 1 is the first study drug day) to 57, Days 3 to 58, etcetera). The double-blind treatment phase was defined as the period between the 1st dosing up until 28 days after the last study drug dose
Time Frame: From first dose of study drug until 28 days after the last dose, as of the data cut-off date of 17 March 2014; median (minimum, maximum) duration of treatment was 168 (14, 449) and 164 (7, 1158) days in each treatment group respectively.
Population: The Intent-to-Treat (ITT) population includes all participants who were randomized to either lenalidomide or placebo.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: 3 placebo capsules by mouth (PO) daily (QD) for at least 168 days until disease progression occurred, intolerable side effects or withdrawal of consent.
- Lenalidomide: Lenalidomide 10 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 60 mL/min for at least 168 days until disease progression, intolerable side effects or withdrawal of consent.
  Lenalidomide 5 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 40 and < 60 mL/min.
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 79 | 160
percentage of participants | 2.5 | 26.9
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Test type: Superiority; p < 0.001, Fisher Exact; p-value is from Fisher's exact test to compare lenalidomide treatment group to placebo group; Risk Ratio (RR) = 10.616, 95% CI 2-sided [2.639 to 42.702]

2. Primary Outcome: Percentage of Participants With a Erythroid Gene Signature Who Achieved RBC Transfusion Independence for ≥ 56 Days as Determined by an Independent Review Committee (IRC)
Description: The percentage of participants who achieved the 56-day RBC TI response was defined as the absence of any RBC transfusions during any consecutive "rolling" 56-day interval within the double-blind treatment phase (ie, Days 2 (Day 1 is the first study drug day) to 57, Days 3 to 58, etcetera). A participant who achieved at least a 56-day RBC-transfusion-independent response was considered a 56-day RBC-TI responder.
Time Frame: as for outcome 1
Population: Analysis population includes ITT participants with an erythroid gene expression signature.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 3 | 14
percentage of participants | 0.0 | 7.1
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Test type: Superiority; p = 1.000, Fisher Exact; p-value is from Fisher's exact test to compare lenalidomide treatment group to placebo group

3. Secondary Outcome: Percentage of Participants Who Achieved RBC Transfusion Independence With a Duration of ≥ 24 Weeks (168 Days) as Determined by the Sponsor
Description: The 168-day RBC-transfusion-independent response was defined as the absence of any RBC transfusion during any consecutive "rolling" 168 days during the treatment period, for example Days 2 (Day 1 is the first study drug day) to 169, Days 3 to 170, Days 4 to 171, etcetera. A responder was defined as a participant who had a ≥ 168 consecutive days of RBC-transfusion-free period after the first dose of study drug in the treatment phase.
Time Frame: as for outcome 1
Population: The ITT population includes all participants who were randomized to either lenalidomide or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 79 | 160
percentage of participants | 0.0 | 17.5
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is from Fisher's exact test to compare the lenalidomide arm to the placebo arm; Risk Ratio (RR) = 0, 95% CI 2-sided [lower limit 0] (NA for risk ratio is due to 0 responder in placebo group.)

4. Secondary Outcome: Kaplan Meier Estimates of Duration of 56-day RBC Transfusion Independence Response as Determined by the Sponsor
Description: The duration of the first 56-day RBC transfusion-independence response was calculated for those who achieved a response and was dependent on whether a subsequent RBC transfusion was given after the transfusion-free period (response):
  * For those who received a subsequent RBC transfusion after the response starts, the duration of response was not censored, and was calculated as response duration = last day of response - first day of response +1 where the last day of response was defined as 1 day before the first RBC transfusion which was given at 56 days or more after the response starts.
  * For those who did not receive a subsequent RBC transfusion after the response started, the end day of the response was censored and duration of the response was calculated as response duration = date of last RBC transfusion assessment - first day of response+ 1. A responder was a participant who had a ≥ 56 consecutive days of RBC-transfusion-free period after the first study drug treatment period
Time Frame: Response was assessed up to the end of treatment; up to the data cut-off date of 17 Mar 2014.
Population: The analysis was conducted only for those participants who achieved a 56-day transfusion independence response according to the sponsor's assessment. Responders in the intent to treat population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 1 | 41
weeks | NA [NA to NA] — Only one placebo participant achieved the response and the response end date was censored | 30.9 [20.7 to 59.1]
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Test type: Superiority; p = 0.639, Log Rank; p-value from log-rank test to compare lenalidomide and placebo

5. Secondary Outcome: Percentage of Participants Who Achieved an Erythroid Response Based on the Modified International Working Group (IWG) 2006 Criteria
Description: A participant was considered as having achieved an erythroid response if the participant either:
  - had a hemoglobin (Hgb) increase ≥1.5 g/dL compared to baseline and confirmed by another central laboratory hemoglobin value at 4 to 8 weeks after the first Hgb measurement that also increased ≥1.5 g/dL. All Hgb values during this time interval must have had a ≥ 1.5 g/dL increase (ie, no central laboratory Hgb increase during this timeframe could be less <1.5 g/dL) OR - had a 50% reduction in the number of the RBC transfusion units over any consecutive 56 days period compared to the baseline transfusion burden.
  The baseline transfusion burden is the number of units over 112 days by the randomization divided by 2. Only transfusions given for a pre-transfusion Hgb value of 9 g/dL or less were used in this response assessment.
Time Frame: as for outcome 1
Population: The ITT population includes all participants who were randomized to either lenalidomide or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 79 | 160
percentage of participants | 30.4 | 38.8
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Test type: Superiority; p = 0.252, Fisher Exact — p-value is from Fisher's exact test to compare the lenalidomide arm to the placebo arm; Risk Ratio (RR) = 1.276, 95% CI 2-sided [0.867 to 1.877]

6. Secondary Outcome: Time to 56-Day RBC-Transfusion-Independent (TI) Response as Determined by the Sponsor
Description: The time to the first 56-day RBC-transfusion-independent response was calculated for participants who achieved a response. The day from the first dose of study drug to the date at which RBC-transfusion-independence starts was achieved and calculated using: Start date of the first response period - the date of the first study drug +1. A responder was defined as a participant who had a ≥ 56 consecutive days of RBC-transfusion-free period after the first dose of study drug in the treatment phase.
Time Frame: From first dose of study drug until 28 days after the last dose of study drug, as of the data cut-off date of 17 March 2014; median (minimum, maximum) duration of treatment was 168 (14, 449) and 164 (7, 1158) days in each treatment group respectively.
Population: The analysis was conducted only for those participants who achieved a 56-day TI response according to the sponsor's assessment. Responders in the intent to treat population.
Measure: Median (Full Range); unit: weeks
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 1 | 41
weeks | 0.3 [0.3 to 0.3] | 10.1 [0.3 to 23.6]

7. Secondary Outcome: Kaplan Meier Estimates for Progression to Acute Myeloid Leukemia (AML)
Description: Progression to AML is part of the natural course of MDS and is a manifestation of disease progression. The time to progress to AML was calculated from the day of randomization to the first day when AML was diagnosed. Participants who died without AML were censored at the date of death. The participants who were lost to follow-up were censored at the last known day when participants did not have AML. Participants who did not progress to AML at the last follow-up contact were censored at the day of the last follow-up contact.
Time Frame: From randomization to final data cut-off date of 03 Jul 2018; median follow up time for progression to AML was 2.3 years (range = 0 to 5.0 years) in the placebo arm and 2.6 years (range = 0 to 6.4 years) in the lenalidomide arm.
Population: ITT population includes all participants who were randomized and received either lenalidomide or placebo. One participant in the placebo arm was diagnosed as having AML before enrollment and was excluded from all analyses of progression to AML.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 78 | 160
years | NA [NA to NA] — Since only a few patients progressed to AML during the observed time frame, median time of progression to AML could not be estimated. | NA [5.2 to NA] — Since only a few patients progressed to AML during the observed time frame, median time of progression to AML could not be estimated.
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Test type: Superiority; p = 0.864, Log Rank — p-value from log-rank test to compare lenalidomide and placebo

8. Secondary Outcome: Kaplan Meier Estimate for Overall Survival (OS)
Description: Overall survival was assessed using the time between randomization and the date of death or date of censoring. Participants who were alive at a data cutoff date and participants who were lost to follow-up were censored at the last date when participants were known to be alive.
Time Frame: From randomization to final data cut-off date of 03 July 2018; maximum survival follow up was 6.4 years
Population: The ITT population includes all participants who were randomized to either lenalidomide or placebo.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 79 | 160
years | 3.0 [2.3 to NA] — Placebo upper limit not estimable. | 3.8 [2.9 to 4.8]
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Test type: Superiority; p = 0.980, Log Rank — p-value from log-rank test to compare lenalidomide and placebo

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: A TEAE was defined as an AE that begins or worsens in intensity of frequency on or after the first dose of study drug through 28 days after last dose of study drug.
  A serious adverse event (SAE) is any:
  * Death;
  * Life-threatening event;
  * Any inpatient hospitalization or prolongation of existing hospitalization;
  * Persistent or significant disability or incapacity;
  * Congenital anomaly or birth defect;
  * Any other important medical event
  The investigator determined the relationship of an AE to study drug based on the timing of the AE relative to drug administration and whether or not other drugs, therapeutic interventions, or underlying conditions could provide a sufficient explanation for the event. The severity of an AE was evaluated by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (Version 3.0) where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death.
Time Frame: From the first dose of study drug through 28 days after discontinuation from the study treatment; up to the final data cut-off date of 03 July 2018; maximum exposure was 2100 days in the lenalidomide arm and 529 days in the placebo arm.
Population: Safety population includes all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: 3 placebo capsules by mouth (PO) daily (QD) for at least 168 days until disease progression occurred or intolerable side effects.
- Lenalidomide: Lenalidomide 10 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 60 mL/min for at least 168 days until disease progression or intolerable side effects.
  Lenalidomide 5 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance between 40 and 60 mL/min.
  .
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 79 | 160
Participants
  At least 1 TEAE | 74 | 160
  ≥ 1 Treatment Related AE (TEAE) | 42 | 144
  ≥ 1 Treatment related TEAE Causing Discontinuation | 3 | 40
  ≥ 1 TEAE Leading to Dose Reduction | 1 | 10
  ≥ 1 TEAE Leading to Dose Interruption | 11 | 89
  ≥ 1 TEAE Leading to Dose Interruption & Reduction | 5 | 68
  ≥ 1 TEAE Leading to Discontinuation of Study Drug | 9 | 51
  ≥ 1 Serious TEAE | 16 | 62
  ≥1 Treatment-Related Serious TEAE | 3 | 25
  ≥1 Serious TEAE Leading to Dose Reduction | 0 | 1
  ≥1 serious TEAE leading to dose interruption | 4 | 21
  ≥1 SAE Causing Dose Interruption & reduction | 1 | 3
  ≥1 Serious TEAE Leading to Stopping of Study Drug | 4 | 24
  ≥1 Grade (GR) 3-4 TEAE | 35 | 139
  ≥ 1 GR 3-4 Related TEAE | 16 | 127
  ≥ 1 GR 3-4 Leading to Dose Reduction | 1 | 8
  ≥ 1 GR 3-4 TEAE Leading to Dose Interruption | 9 | 80
  ≥ 1 GR 3-4 TEAE dose Interruption &reduction | 4 | 64
  ≥ 1 GR 3-4 TEAE Leading to Stopping of Study Med | 6 | 41
  ≥ 1 GR 5 TEAE | 2 | 6
  ≥1 GR Treatment Related 5 TEAE | 1 | 3

10. Secondary Outcome: Compliance Rates Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) From Baseline to Week 48
Description: The European Organization for Research and Treatment of Cancer QOL Questionnaire for Patients with Cancer (EORTC QLQ-C30) was a 30-item oncology-specific questionnaire. The questionnaire was developed to assess the quality of life of cancer patients. It contains 30 questions, 24 of which form 9 multi-item scales representing various aspects of HRQOL: 1 global scale, 5 functional scales (Physical, Role, Emotional, Cognitive and Social), and 3 symptom scales (Fatigue, Pain, and Nausea). The remaining 6 items are intended to be mono-item scales describing relevant cancer-oriented symptoms (dyspnea, insomnia, appetite, constipation, diarrhea, financial difficulties). Subscale scores are transformed to a 0 to 100 scale, with higher scores on functional scales indicating better function and higher score on symptom scales indicating worse symptoms. A participant was considered compliant at a visit if at least 15 out of the QLQ-C30 items in the questionnaire were checked.
Time Frame: Baseline, Week 12, (±3 days), Week 24, (±3 days), Week 36, (±3 days), and Week 48 (±3 days); up to data cut-off of 17 Mar 2014
Population: Analyses were performed based on the Health Related Quality of Life (HRQoL) evaluable population, defined as all randomized participants who completed the baseline assessment and at least one post-baseline assessment for the intent to treat population. Data is available up to Week 48 due to small sample after that.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 79 | 160
percentage of participants
  Baseline | 88.6 | 90
  Week 12 | 78.5 | 83.8
  Week 24 | 80.6 | 85.8
  Week 36 | 100 | 80.5
  Week 48 | 50 | 71.9
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Baseline; Test type: Superiority; p = 0.823, Fisher Exact; The p-values are calculated based on the Fisher exact test
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 12 (±3 days); Test type: Superiority; p = 0.371, Fisher Exact; The p-values are calculated based on the Fisher exact test
Statistical Analysis 3: Comparison: Placebo vs Lenalidomide; Week 24 (±3 days); Test type: Superiority; p = 0.391, Fisher Exact; The p-values are calculated based on the Fisher exact test
Statistical Analysis 4: Comparison: Placebo vs Lenalidomide; Week 36 (±3 days); Test type: Superiority; p = 1.000, Fisher Exact; The p-values are calculated based on the Fisher exact test
Statistical Analysis 5: Comparison: Placebo vs Lenalidomide; Week 48 (±3 days); Test type: Superiority; p = 0.508, Fisher Exact; The p-values are calculated based on the Fisher exact test

11. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Fatigue Domain at Week 12 and 24
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Fatigue Scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate reduction in fatigue (i.e. improvement in symptom) and positive values indicate increases in fatigue (i.e. worsening of symptom).
Time Frame: Baseline and Week 12, ±3 days and Week 24, ±3 days
Population: Analyses were performed based on the HRQoL evaluable population, defined as all randomized participants who completed the baseline assessment and at least one post-baseline assessment for the intent to treat population. Only those with available data at baseline and each time point are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lenalidomide: .Lenalidomide 10 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 60 mL/min for at least 168 days until disease progression, intolerable side effects or withdrawal of consent.
  Lenalidomide 5 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 40 and < 60 mL/min.
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
units on a scale
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 0.6 (17.53) | 2.4 (28.26)
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | 7.6 (20.74) | -1.5 (26.42)
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.323, ANOVA; P-value from ANOVA comparison for change from baseline between lenalidomide and placebo adjusted with baseline score
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.071, ANOVA — P-value from ANOVA comparison for change from baseline between lenalidomide and placebo adjusted with baseline score

12. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Dyspnea Domain at Week 12 and 24
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Dyspnea scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate decreased dyspnea (i.e. improvement in symptom) and positive values indicate increased dyspnea (i.e. worsening of symptom).
Time Frame: Baseline and Week 12, ±3 days and Week 24, ±3 days
Population: Analyses were performed based on the Health Related Quality of Life (HRQoL) evaluable population, defined as all randomized participants who completed the baseline assessment and at least one post-baseline assessment for the intent to treat population. Only those with available data at baseline and each time point are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: 3 placebo capsules by mouth (PO) daily (QD) for at least 168 days until disease progression occurred or intolerable side effects or withdrawal of consent.
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
units on a scale
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 0.6 (28.06) | 2.2 (29.92)
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | 4.3 (26.57) | 1.2 (26.26)
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.760, ANOVA — P-value from ANOVA comparison for change from baseline between lenalidomide and placebo adjusted with baseline score
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.251, ANOVA — P-value from ANOVA comparison for change from baseline between lenalidomide and placebo adjusted with baseline score

13. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Physical Functioning Domain at Week 12 and 24
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Physical Functioning Scale was scored between 0 and 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Baseline and Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
units on a scale
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | -1.4 (15.76) | -2.1 (18.09)
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | -5.7 (14.84) | -0.4 (18.19)
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.424, ANOVA — P-value from ANOVA comparison for change from baseline between lenalidomide and placebo adjusted with baseline score
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.116, ANOVA — P-value from ANOVA comparison for change from baseline between lenalidomide and placebo adjusted with baseline score

14. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Global Health Status/Quality of Life (QOL) Domain at Week 12 and 24
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Global Health Status/QOL scale was scored between 0 and 100, with a high score indicating better Global Health Status/QOL. Negative change from Baseline values indicate deterioration in Global Health Status/QOL and positive values indicate improvement.
Time Frame: Baseline and Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
units on a scale
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | -2.1 (20.18) | -1.4 (24.35)
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | -4.1 (20.25) | -2.4 (27.87)
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.746, ANOVA — P-value from ANOVA comparison for change from baseline between lenalidomide and placebo adjusted with baseline score
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Test type: Superiority; p = 0.460, ANOVA — P-value from ANOVA comparison for change from baseline between lenalidomide and placebo adjusted with baseline score

15. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Emotional Functioning Domain at Week 12 and 24
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Emotional Functioning Domain was scored between 0 and 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Baseline and Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lenalidomide: Lenalidomide 10 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 60 mL/min for at least 168 days until disease progression, intolerable side effects or withdrawal of consent.
  Lenalidomide 5 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 40 and < 60 mL/min.
  .
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
units on a scale
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 1.2 (18.70) | -1.4 (22.39)
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | -7.1 (20.78) | 0.8 (20.06)
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.265, ANOVA — P-value from ANOVA comparison for change from baseline between lenalidomide and placebo adjusted with baseline score
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.047, ANOVA — 3]: P-value from ANOVA comparison for change from baseline between lenalidomide and placebo adjusted with baseline score

16. Secondary Outcome: Mean Change From Baseline in Fatigue Domain Associated With the EORTC QLQ-C-30 Scale at Week 12 and Week 24
Description: The European Organization for Research and Treatment of Cancer QOL Questionnaire for Patients with Cancer (EORTC QLQ-C30) was a 30-item oncology-specific questionnaire. The questionnaire was developed to assess the quality of life of cancer patients. It contains 30 questions, 24 of which form 9 multi-item scales representing various aspects of HRQOL: 1 global scale, 5 functional scales (Physical, Role, Emotional, Cognitive and Social), and 3 symptom scales (Fatigue, Pain, and Nausea). The remaining 6 items are intended to be mono-item scales describing relevant cancer-oriented symptoms (dyspnea, insomnia, appetite, constipation, diarrhea, financial difficulties). The EORTC QLQ-C30 Fatigue Scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate reduction in fatigue (i.e. improvement in symptom) and positive values indicate increases in fatigue (i.e. worsening of symptom).
Time Frame: Baseline, Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
units on a scale
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | -0.464 [-6.562 to 5.635] | 3.497 [-0.631 to 7.624]
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | 7.376 [0.990 to 13.762] | 0.196 [-4.505 to 4.897]
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.2909, t-test, 2 sided — P-value is based on a two-sample t-test comparing the difference between treatments
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.0759, t-test, 2 sided — P-value is based on a two-sample t-test comparing the difference between treatments

17. Secondary Outcome: Mean Change From Baseline in the Dyspnea Domain Associated With the EORTC QLQ-C-30 Scale at Week 12 and Week 24
Description: as for outcome 12
Time Frame: Baseline, Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
units on a scale
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 1.696 [-5.313 to 8.706] | 3.374 [-1.369 to 8.117]
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | 5.998 [-1.174 to 13.171] | -0.206 [-5.557 to 5.146]
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.6957, t-test, 2 sided — P-value is based on a two-sample t-test comparing the difference between treatments
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.1729, t-test, 2 sided — P-value is based on a two-sample t-test comparing the difference between treatments

18. Secondary Outcome: Mean Change From Baseline in the Physical Functioning Domain Associated With the EORTC QLQ-C-30 Scale at Week 12 and Week 24
Description: The European Organization for Research and Treatment of Cancer QOL Questionnaire for Patients with Cancer (EORTC QLQ-C30) was a 30-item oncology-specific questionnaire. The questionnaire was developed to assess the quality of life of cancer patients. It contains 30 questions, 24 of which form 9 multi-item scales representing various aspects of HRQOL: 1 global scale, 5 functional scales (Physical, Role, Emotional, Cognitive and Social), and 3 symptom scales (Fatigue, Pain, and Nausea). The remaining 6 items are intended to be mono-item scales describing relevant cancer-oriented symptoms (dyspnea, insomnia, appetite, constipation, diarrhea, financial difficulties). The EORTC QLQ-C30 Physical Functioning was scored between 0 and 100, with a high score indicating better Global Health Status/QOL. Negative change from Baseline values indicate deterioration in Global Health Status/QOL and positive values indicate improvement.
Time Frame: Baseline, Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
units on a scale
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 0.732 [-4.939 to 3.475] | -2.919 [-5.768 to -0.071]
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | -5.451 [-10.046 to -0.85] | -1.484 [-4.861 to 1.892]
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.3975, t-test, 2 sided; P-value is based on a two-sample t-test comparing the difference between treatments
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.1714, t-test, 2 sided — P-value is based on a two-sample t-test comparing the difference between treatments

19. Secondary Outcome: Mean Change From Baseline in the Global Health Status/QoL Domain Associated With the EORTC QLQ-C-30 Scale at Week 12 and Week 24
Description: The European Organization for Research and Treatment of Cancer QOL Questionnaire for Patients with Cancer (EORTC QLQ-C30) was a 30-item oncology-specific questionnaire. The questionnaire was developed to assess the quality of life of cancer patients. It contains 30 questions, 24 of which form 9 multi-item scales representing various aspects of HRQOL: 1 global scale, 5 functional scales (Physical, Role, Emotional, Cognitive and Social), and 3 symptom scales (Fatigue, Pain, and Nausea). The remaining 6 items are intended to be mono-item scales describing relevant cancer-oriented symptoms (dyspnea, insomnia, appetite, constipation, diarrhea, financial difficulties). The EORTC QLQ-C30 Global Health Status/QOL scale was scored between 0 and 100, with a high score indicating better Global Health Status/QOL. Negative change from Baseline values indicate deterioration in Global Health Status/QOL and positive values indicate improvement.
Time Frame: Baseline, Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
units on a scale
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | -1.201 [-6.401 to 3.999] | -2.690 [-6.211 to 0.831]
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | -4.502 [-10.330 to 1.326] | -2.441 [-6.761 to 1.880]
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.6408, t-test, 2 sided — P-value is based on a two-sample t-test comparing the difference between treatments
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.5750, t-test, 2 sided — P-value is based on a two-sample t-test comparing the difference between treatments

20. Secondary Outcome: Mean Change From Baseline in the Emotional Functioning Domain Associated With the EORTC QLQ-C30 Scale at Weeks 12 and 24
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Emotional Functioning Scale is scored between 0 and 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Baseline, Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
units on a scale
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 1.458 [-3.621 to 6.536] | -1.876 [-5.307 to 1.556]
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | -6.746 [-12.228 to -1.26] | -1.129 [-5.174 to 2.917]
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.2848, t-test, 2 sided; P-value is based on a two-sample t-test comparing the difference between treatments
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.1053, t-test, 1 sided — P-value is based on a two-sample t-test comparing the difference between treatments

21. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvement in QOL (EORTC QLQ-C-30 Scale) From Baseline in Fatigue Domain at Weeks 12 and 24
Description: The European Organization for Research and Treatment of Cancer QOL Questionnaire for Patients with Cancer (EORTC QLQ-C30) was a 30-item oncology-specific questionnaire. The questionnaire was developed to assess the quality of life of cancer patients. It contains 30 questions, 24 of which form 9 multi-item scales representing various aspects of HRQOL: 1 global scale, 5 functional scales (Physical, Role, Emotional, Cognitive and Social), and 3 symptom scales (Fatigue, Pain, and Nausea). The remaining 6 items are intended to be mono-item scales describing relevant cancer-oriented symptoms (dyspnea, insomnia, appetite, constipation, diarrhea, financial difficulties). Subscale scores are transformed to a 0 to 100 scale, with higher scores on functional scales indicating better function and higher score on symptom scales indicating worse symptoms. Improvement means at least 10 points better compared to baseline
Time Frame: Baseline, Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
percentage of participants
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 30.4 | 39.3
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | 29.8 | 38.6
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.042, Fisher Exact — The P-values are calculated based on Fisher exact test
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.448, Fisher Exact — The P-values are calculated based on Fisher exact test

22. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvement in HRQOL Associated With the EORTC QLQ-C-30 Scale From Baseline in the Dyspnea Domain at Weeks 12 and 24
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Dyspnea scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate decreased dyspnea (i.e. improvement in symptom) and positive values indicate increased dyspnea (i.e. worsening of symptom). Improvement means at least 10 points better compared to baseline.
Time Frame: Baseline, Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
percentage of participants
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 19.6 | 21.3
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | 12.8 | 20.5
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.825, Fisher Exact — The P-values are calculated based on Fisher exact test
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.568, Fisher Exact — The P-values are calculated based on Fisher exact test

23. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvement in HRQOL Associated With the EORTC QLQ-C-30 Scale From Baseline Within the Physical Functioning Domain at Weeks 12 and 24
Description: The European Organization for Research and Treatment of Cancer QOL Questionnaire for Patients with Cancer (EORTC QLQ-C30) was a 30-item oncology-specific questionnaire. The questionnaire was developed to assess the quality of life of cancer patients. It contains 30 questions, 24 of which form 9 multi-item scales representing various aspects of HRQOL: 1 global scale, 5 functional scales (Physical, Role, Emotional, Cognitive and Social), and 3 symptom scales (Fatigue, Pain, and Nausea). The remaining 6 items are intended to be mono-item scales describing relevant cancer-oriented symptoms (dyspnea, insomnia, appetite, constipation, diarrhea, financial difficulties). Subscale scores are transformed to a 0 to 100 scale, with higher scores on functional scales indicating better function and higher score on symptom scales indicating worse symptoms. A change of at least 10 points on the standardized domain scores was required for it to be considered clinically meaningful.
Time Frame: Baseline, Week 12, ±3 days and Week 24, ±3 days
Population: Analyses were performed based on the HRQoL evaluable population, defined as all randomized participants who completed the baseline assessment and at least one post-baseline assessment with the EORTC QLQ-C-30. Only those with available data at baseline and each time point are included.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
percentage of participants
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 26.8 | 16.4
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | 12.8 | 24.1
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.119, Fisher Exact — The P-values are calculated based on Fisher exact test
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.172, Fisher Exact — The P-values are calculated based on Fisher exact test

24. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvement in HRQOL Associated With the EORTC QLQ-C-30 Scale From Baseline in the Global Health Status/QOL Domain at Weeks 12 and 24
Description: as for outcome 23
Time Frame: Baseline, Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
percentage of participants
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 19.6 | 22.1
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | 14.9 | 26.5
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.792, Fisher Exact — The P-values were calculated based on Fisher exact test
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.279, Fisher Exact — The P-values are calculated based on Fisher exact test

25. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvement in HRQOL Associated With the EORTC QLQ-C-30 Scale From Baseline in the Emotional Functioning Domain at Weeks 12 and 24
Description: as for outcome 15
Time Frame: Baseline, Week 12, ±3 days and Week 24, ±3 days
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 58 | 131
percentage of participants
  Week 12: number analyzed (Participants) | 56 | 122
  Week 12 | 25.0 | 20.5
  Week 24: number analyzed (Participants) | 47 | 83
  Week 24 | 17.0 | 21.7
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Week 12; Test type: Superiority; p = 0.476, Fisher Exact — The P-values are calculated based on Fisher exact test
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide; Week 24; Test type: Superiority; p = 0.052, Fisher Exact — The P-values are calculated based on Fisher exact test

26. Post Hoc Outcome: Percentage of Participants Who Achieved an Erythroid Response Based on Original IWG 2006 Criteria
Description: A participant was considered as having achieved an erythroid response when:
  - a Hgb increase ≥1.5 g/dL compared to baseline and confirmed by another central laboratory hemoglobin value at 4 to 8 weeks after the first Hgb measurement that had also increased ≥1.5 g/dL for at least 8 weeks. All Hgb values during this time interval must have had a ≥ 1.5 g/dL increase (ie, no central laboratory Hgb increase during this timeframe can be less than a 1.5 g/dL) OR - had an absolute reduction of 4 RBC transfusion units over any consecutive 56 days period compared to the baseline transfusion burden.
  The baseline transfusion burden is the number of units over the 112 days prior to randomization divided by 2. Only transfusions given for a pre-transfusion Hgb value of 9.5 g/dL or less may be used in this response assessment.
Time Frame: as for outcome 1
Population: Intent to treat population includes all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 79 | 160
percentage of participants | 20.3 | 35.6
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide; Test type: Superiority; p = 0.017, Fisher Exact — p-value is from Fisher's exact test to compare lenalidomide treatment group to placebo group; Risk Ratio (RR) = 1.759, 95% CI 2-sided [1.083 to 2.856]

27. Secondary Outcome: Healthcare Resource Utilization (HRU): Rate of Inpatient Hospitalizations Related to Adverse Events Per Person Year
Description: Hospitalizations due to adverse events exclude those for transfusions, elective procedures or protocol-driven procedures. HRU was defined as any consumption of healthcare resources directly or indirectly related to the treatment of the patient.
Time Frame: as for outcome 1
Population: Safety population includes all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Hospitalizations per person-years
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 79 | 160
Hospitalizations per person-years | 0.47 [0.3 to 0.75] | 0.77 [0.62 to 0.96]

28. Secondary Outcome: Healthcare Resource Utilization (HRU): Duration of Hospitalizations Due to Adverse Events
Description: as for outcome 27
Time Frame: as for outcome 1
Population: Participants with at least one hospitalization.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 14 | 57
Days | 9.0 [1.0 to 66.0] | 11.0 [1.0 to 76.0]

29. Secondary Outcome: Healthcare Resource Utilization (HRU): Number of Days of Hospitalization Due to Adverse Events Per Person-Years
Description: as for outcome 27
Time Frame: as for outcome 1
Population: Safety population includes all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Days per person-years
Arm/Group | Placebo | Lenalidomide
Number analyzed (Participants) | 79 | 160
Days per person-years | 6.37 [4.64 to 8.74] | 8.92 [7.35 to 10.82]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through 28 days after last dose; up to the final data cut-off date of 03 July 2018; maximum exposure was 2100 days in the lenalidomide treatment group and 529 days in the placebo group
Description: Second primary malignancies were monitored as events of interest and reported as serious adverse events for at least 5 years from randomization unless the participants withdrew consent from the study, died or were lost to follow-up.
Groups:
- Placebo: Participants received 3 placebo capsules by mouth QD for at least 168 days until disease progression occurred, intolerable side effects or withdrawal of consent
- Lenalidomide: Participants received lenalidomide 10 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance ≥ 60 mL/min for at least 168 days until disease progression or intolerable side effects. Lenalidomide 5 mg PO daily plus 2 placebo capsules for participants with a creatinine clearance between 40 and 60 mL/min.
Arm/Group | Placebo | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 43/79 | 94/160
Serious Adverse Events (participants affected / at risk) | 16/79 | 62/160
Other Adverse Events (participants affected / at risk) | 70/79 | 154/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Lenalidomide (N=160)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 5
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 3
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 1
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 2 | 3
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 2
TACHYARRHYTHMIA (Cardiac disorders) | 0 | 1
CATARACT (Eye disorders) | 0 | 1
ULCERATIVE KERATITIS (Eye disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
ASCITES (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS NECROTISING (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
DISUSE SYNDROME (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 2
MALAISE (General disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
PYREXIA (General disorders) | 0 | 1
SUDDEN DEATH (General disorders) | 0 | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1
ATYPICAL PNEUMONIA (Infections and infestations) | 0 | 1
BRONCHITIS (Infections and infestations) | 2 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 2
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 3
PNEUMONIA (Infections and infestations) | 2 | 10
PNEUMONIA VIRAL (Infections and infestations) | 0 | 1
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
TOOTH ABSCESS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CHRONIC MYELOMONOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG SQUAMOUS CELL CARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF THE TONGUE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1
DYSKINESIA (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 2
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 3
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
NEURODERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 2
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Lenalidomide (N=160)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 8
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 22
NEUTROPENIA (Blood and lymphatic system disorders) | 9 | 102
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 | 66
CONJUNCTIVITIS (Eye disorders) | 0 | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 10
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 | 12
CONSTIPATION (Gastrointestinal disorders) | 9 | 36
DIARRHOEA (Gastrointestinal disorders) | 18 | 69
DYSPEPSIA (Gastrointestinal disorders) | 2 | 8
NAUSEA (Gastrointestinal disorders) | 12 | 19
VOMITING (Gastrointestinal disorders) | 5 | 13
ASTHENIA (General disorders) | 13 | 38
FATIGUE (General disorders) | 9 | 36
OEDEMA PERIPHERAL (General disorders) | 14 | 35
PYREXIA (General disorders) | 6 | 20
INFLUENZA (Infections and infestations) | 2 | 10
NASOPHARYNGITIS (Infections and infestations) | 9 | 19
PNEUMONIA (Infections and infestations) | 4 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 4
URINARY TRACT INFECTION (Infections and infestations) | 6 | 9
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 15
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 13
SERUM FERRITIN INCREASED (Investigations) | 4 | 1
WEIGHT DECREASED (Investigations) | 2 | 17
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 | 19
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 10
IRON OVERLOAD (Metabolism and nutrition disorders) | 4 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 | 14
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 | 16
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 19
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 8
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 18
DIZZINESS (Nervous system disorders) | 9 | 13
HEADACHE (Nervous system disorders) | 8 | 9
INSOMNIA (Psychiatric disorders) | 7 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 17
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 | 15
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 10
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 12
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 3 | 8
PRURITUS (Skin and subcutaneous tissue disorders) | 9 | 30
RASH (Skin and subcutaneous tissue disorders) | 4 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 12 months since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.